CLINICAL TRIAL: NCT03854058
Title: Multimodal Measurement of Respiratory Muscle Strength by Using Volitional and Non-volitional Tests in Patients With Obesity Hypoventilation Syndrome (OHS), Obesity-associated Hypoventilation and OHS-Risk-Patients to Evaluate Pathophysiological Determinants and Predictors for the Presence of a Sleep-related Hypoventilation Requiring Treatment in Obese Patients
Brief Title: Respiratory Muscle Strength in Patients With Obesity Hypoventilation Syndrome (OHS) or With a Precursor of the Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_18-340
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Spirometry; Polysomnography; Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHS or elevated OHS-risk (stages 0-IV): stage 0: OHS-risk (OSA / no hypercapnia)
  stage I: obesity associated hypoventilation (intermittent hypercapnia during sleep, arterial carbon dioxide partial pressure (PaCO2) or transcutaneous carbon dioxide partial pressure (PtcCO2) morning ~ evening), bicarbonate < 27 mmol/L awake)
  stage II: obesity associated hypoventilation (intermittent hypercapnia during sleep, PaCO2 or PtcCO2 morning > evening, bicarbonate ≥ 27 mmol/L awake)
  stage III: OHS (hypercapnia, carbon dioxide partial pressure (PCO2) > 45 mmHg awake)
  stage IV: OHS with end organ damage (hypercapnia , PCO2 > 45 mmHg awake, cardiometabolic comorbidities)
  diagnostic tests: magnetic phrenic nerve stimulation, diaphragmatic ultrasound
  Interventions: Diagnostic Test: magnetic phrenic nerve stimulation

INTERVENTIONS:
Diagnostic Test: magnetic phrenic nerve stimulation — cervical and cortical stimulation of N. Vagus
  Other Names: diaphragmatic ultrasound; spirometry; Sleep-studies; capnography

SUMMARY:
Using an extensive set of both volitional and non-volitional tests of respiratory muscle function and strength it is the aim of this study to

* identify potential determinants for the development of obesity hypoventilation
* to identify predictors for the presence of a sleep-related hypoventilation requiring treatment in obese patients

ELIGIBILITY:
Inclusion Criteria:

* patients with BMI > 30 and obesity-associated hypoventilation stages I - IV
* patients with BMI > 30 and elevated OHS-risk (= obstructive sleep apnea without hypercapnia)
* age:18-80 years
* capacity to consent

Exclusion Criteria:

* any other disease, that causes ventilatory insufficiency
* pacemaker, defibrillators or device for deep brain or vagus nerve stimulation
* esophagitis, Barrett-esophagus, esophageal cancer
* acute gastritis and ulcera ventriculi
* epilepsy
* any medical, psychological or other condition impairing the patient's ability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OHS or OHS-risk
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Carbon dioxide rebreathing test | 1 day
  minute volumen (L/min)
transdiaphragmatic pressure (non-volitional) | 1 day
  difference between intraesophageal and intragastral pressure after posterior magnetic stimulation of the phrenic nerves
peripheral nervous system (non-volitional) | 1 day
  electroneurography after posterior magnetic stimulation of the phrenic nerves
diaphragmal ultrasound - excursion (non-volitional) | 1 day
  excursion of the diaphragm
diaphragmal ultrasound - thickness (non-volitional) | 1 day
  thickness of the diaphragm
P0.1 (volitional) | 1 day
  mouth occlusion pressure (kPa)
PImax (volitional) | 1 day
  maximal inspiratory mouth pressure (kPa)

SECONDARY OUTCOMES:
Comparison of PImax and transdiaphragmatic pressure | 1 day
  Correlation between PImax and transdiaphragmatic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Institut für Pneumologie an der Universität zu Köln / Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No